CLINICAL TRIAL: NCT02696005
Title: Hormone KLOTHO Level in Heart Failure Patients That Participate in Rehabilitation Programme
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 109-15-BNZ
Record Dates: First submitted 2015-12-30; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: 15 patients who will continue participation in Exercise- Based Cardiac Rehabilitation Programme after completion initial 3-months period.
  Interventions: Other: Exercise- Based Cardiac Rehabilitation Programme
- Group II: 15 patients who will stop participation in Exercise- Based Cardiac Rehabilitation Programme after the initial 3-months period.
  Interventions: Other: Exercise- Based Cardiac Rehabilitation Programme

INTERVENTIONS:
Other: Exercise- Based Cardiac Rehabilitation Programme — Exercise- Based Cardiac Rehabilitation Programme for patients suffering from Heart Failure.
  Other Names: Rehabilitation Programme

SUMMARY:
30 patients suffering from Heart Failure with Ejection Fraction less than 40% start Cardiac Rehabilitation Programme, serum KLOTHO Hormone level and other labs and Echo measurements will be taken on the first visit.

After completion of 3-month Rehabilitation Programme the second set of labs and Echo measurements will be taken.

Than participants will be divided for 2 groups: the patients who wish to continue Rehabilitation programme for additional 3-month period and the second group that prefer to stop Rehabilitation programme after completion of the first 3 month period.

For both groups additional set of labs will be taken this time and at the end of the study.

The Aim of the study: to investigate association between serum KLOTHO level, physical activity and possible correlation with laboratory and echocardiographic parameters in cohort of Heart Failure patients.

DETAILED DESCRIPTION:
30 patients, age range older than 18 years old suffering from Heart Failure, Functional capacity II-III and echocardiographic evidence of Left Ventricular Ejection Fraction less than 40% beginning Cardiac Rehabilitation Programme. Following recruitment of patients to the study each one will undergo serum KLOTHO Hormone level assessment along with kidney functions, N terminal -Pro B-Type Natriuretic Peptide hormone activity and Echo measurements .

After completion of 3-months Exercise based Rehabilitation Programme set at 70-80% of maximal individual exercise capacity,a second identical set of lab tests and Echo measurements will be performed.

After than participants will be divided into 2 groups: Group I will comprise patients who wish to continue Rehabilitation programme for additional 3-months period and the Group II those who will stop Exercise Rehabilitation programme following completion of the first 3 months.

Both groups will undergo additional set of lab tests at this six-months-point. Except for the primary and secondary end-points all possible correlations between serum KLOTHO level and age, sex, Ejection Fraction, functional capacity, N terminal -Pro B-Type Natriuretic Peptide hormone activity hormone level and kidney function indices will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Patients ≥ than 18 years
3. Ejection Fraction ≤ than 40 %

Exclusion Criteria:

1. Myocardial Infarction ≤ than 1.5 month before inclusion
2. Renal failure with Creatinine ≥ 1.5 mg/dl
3. Known Inflammatory condition.
4. Patient taking Calcium Supplement,Vitamin D or pyrophosphate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients suffering from Heart Failure and beginning Rehabilitation Programme
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Serum Klotho hormone level | "Baseline", "3 months" and "6 months"
  Change in serum Klotho level between "Baseline", "3 months" and "6 months" visits

SECONDARY OUTCOMES:
Incidence of Hospital Readmissions in patients with different serum level of KLOTHO | "3 months" and "6 months" and "1 Year"

CONTACTS AND LOCATIONS:
Overall Officials: Eugeny Radzishevsky, MD, Principal Investigator — Bnai Zion Medical Center- Ministry of Health, Israel

IPD SHARING:
Plan to Share IPD: No